CLINICAL TRIAL: NCT05093101
Title: The Prognostic Value of Serum Biomarkers in Osteosarcoma
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Costantino Errani, Principal Investigator, Istituto Ortopedico Rizzoli
Other Study IDs: ProOsteo
Record Dates: First submitted 2021-10-12; First posted 2021-10-26 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2021-10

CONDITIONS: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: case series review of clinical data — Extraction of pre-surgical and chemotherapy blood test laboratory data and clinical and instrumental data related to patient history from digitized medical records and analysis

SUMMARY:
Observational retrospective cohort study using laboratory data of blood tests prior to surgical and chemotherapy treatment and other histologic, clinical, and instrumental data related to patient history from digitized medical records and analysis of the same as predictors of outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Osteosarcoma diagnosed at the Pathological Anatomy of the Rizzoli Orthopaedic Institute in Bologna;
* Minimum 2-year follow-up period;
* Medical records, complete blood work and instrumental examinations, regular follow-up;
* Patients with age ≥ 2 years;

Exclusion Criteria:

* Patients with osteosarcoma who have received medical treatment (surgery, radiotherapy or chemotherapy) in other hospitals prior to admission to our Institute

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: pazients with osteosarcoma from 01-01-2000 to 31-12-2020
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Evaluation of 5-year survival | 5 years
  Evaluation of 5-year survival in relation to histologic, laboratory, clinical, and instrumental prognostic factors

SECONDARY OUTCOMES:
Evaluation of the rate of local recurrence | 5 years
  Evaluation of the rate of local recurrence and distant metastasis in relation to histological, laboratory, clinical, and instrumental prognostic factors.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Itituto Ortopedico Rizzoli, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nakamura T, Grimer RJ, Gaston CL, Watanuki M, Sudo A, Jeys L. The prognostic value of the serum level of C-reactive protein for the survival of patients with a primary sarcoma of bone. Bone Joint J. 2013 Mar;95-B(3):411-8. doi: 10.1302/0301-620X.95B3.30344. PMID 23450030
- [Result] Li YJ, Yang X, Zhang WB, Yi C, Wang F, Li P. Clinical implications of six inflammatory biomarkers as prognostic indicators in Ewing sarcoma. Cancer Manag Res. 2017 Sep 28;9:443-451. doi: 10.2147/CMAR.S146827. eCollection 2017. PMID 29033609
- [Result] Aggerholm-Pedersen N, Maretty-Kongstad K, Keller J, Baerentzen S, Safwat A. The Prognostic Value of Serum Biomarkers in Localized Bone Sarcoma. Transl Oncol. 2016 Aug;9(4):322-8. doi: 10.1016/j.tranon.2016.05.006. PMID 27567955
- [Derived] Basoli S, Cosentino M, Traversari M, Manfrini M, Tsukamoto S, Mavrogenis AF, Bordini B, Donati DM, Errani C. The Prognostic Value of Serum Biomarkers for Survival of Children with Osteosarcoma of the Extremities. Curr Oncol. 2023 Jul 24;30(7):7043-7054. doi: 10.3390/curroncol30070511. PMID 37504371